CLINICAL TRIAL: NCT00458445
Title: A Phase IIIb Study to Evaluate the Efficacy and Time Course of Treatment With SPD465 Compared to Placebo on Simulated Driving Safety and Performance in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: A Study of SPD465 in Young Adult Drivers With Attention-Deficit Hyperactivity Disorder (ADHD) Using Driving Simulators
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was stopped by the sponsor before enrollment based on a non-safety related corporate decision.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SPD465-311
Record Dates: First submitted 2007-04-02; First posted 2007-04-10 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention-Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- SPD465 then Placebo (Experimental)
  Interventions: Drug: SPD465; Other: Placebo
- Placebo then SPD465 (Experimental)
  Interventions: Drug: SPD465; Other: Placebo

INTERVENTIONS:
Drug: SPD465
Other: Placebo — Placebo is a material that may look similar to SPD465, however, contains no active drug.

SUMMARY:
The purpose of this study is to determine whether SPD465 is safe and effective in the treatment of ADHD in young adult drivers after a duration of 16 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a valid driver's license with a minimum of 3 years of driving experience.
2. Subject reports daily driving activity.
3. Subject is fluent in English.
4. Subject must be male or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol.
5. Subject must have a satisfactory medical assessment with no clinically significant or relevant abnormalities
6. Subject meets DSM-IV-TR criteria for a primary diagnosis of ADHD) established by a comprehensive psychiatric evaluation that reviews DSM-IV-TR criteria

Exclusion criteria:

1. Subject is significantly underweight or morbidly obese.
2. Subject has a controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as Post Traumatic Stress Disorder (PTSD), psychosis, bipolar illness, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder or other symptomatic manifestations that, in the opinion of the examining Physician, will contraindicate SPD465 treatment or confound efficacy or safety assessments.
3. Subject with a lifetime history of psychosis or bipolar disorder.
4. Subject with any concurrent chronic or acute illness or unstable medical condition, either treated or untreated.
5. Subject with a history of mental retardation or a severe learning disability.
6. Subject is naïve to ADHD treatment with methylphenidate or amphetamine.
7. Subject has a history of glaucoma or narrow angle glaucoma.
8. Subject has a history of seizure (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or family history of Tourette's Disorder.
9. Subject has known cardiac structural abnormalities as well as any other condition that may affect cardiac performance.
10. Subject has clinically significant ECG or laboratory abnormalities at Screening or Baseline.
11. Subject has a history of hypertension or has a resting sitting systolic blood pressure >139mmHg or diastolic blood pressure >89mmHg10.
12. Subject has used any psychoactive prescription medication or over-the-counter (OTC) medication requiring more than a 28-day washout. Hormonal contraceptives are acceptable.
13. Subject has a documented allergy, intolerance, or documented history of non-responsivity to amphetamine.
14. Subject currently has (or had a history within the last 6 months) a substance use disorder (excluding nicotine).
15. Subject has taken another investigational drug or taken part in a clinical trial within the last 30 days prior to Screening.
16. Female subject is pregnant or lactating.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04-30 (Actual); Primary Completion 2007-06-15 (Actual); Study Completion 2007-06-15 (Actual)

PRIMARY OUTCOMES:
Simulated Driver Safety (DS) Score averaged over 3 driving assessments at one interim and one final visit. | Interim visit = Week 3; Final visit = Week 7.

SECONDARY OUTCOMES:
Interim & final visits: Attention-Deficit Hyperactivity Disorder Rating Scale - 4th Edition (ADHD-RS-IV) | Interim visit = Week 3; Final visit = Week 7.
Interim & final visits: Clinical Global Impressions of Improvement (CGI-I) | Interim visit = Week 3; Final visit = Week 7.
Interim & final visits: Self-Rating of Simulated Driver Safety (DS) Performance Questionnaire | Post DS Testing - Interim visit = Week 3; Post DS Testing - Final visit = Week 7.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Meridien Research, Tampa, Florida, United States